CLINICAL TRIAL: NCT05080114
Title: A Multimodal Concept for Vaginal Cuff Closure by Modification of the Bakay Technique in Total Laparoscopic Hysterectomy: A Randomized Clinical Study
Brief Title: Vaginal Cuff Closure by Modification of the Bakay Technique in Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Uzeyir Kalkan, Principal Investigator, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMU KAEK 2018/22
Record Dates: First submitted 2021-10-02; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Hysterectomy; Surgery; Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified technique (MT) (Experimental): All the steps of the laparoscopic hysterectomy were performed according to conventional standard technique until the colpotomy step. Instead, the modified Bakay technique was used for later on.
  Interventions: Procedure: Modified Bakay technique (MT)
- Standard technique (ST) (Active Comparator): The conventional standard total laparoscopic hysterectomy technique was used in this control group.
  Interventions: Procedure: Standard technique (ST)

INTERVENTIONS:
Procedure: Modified Bakay technique (MT) — The conventional standard technique for laparoscopic hysterectomy was followed until the colpotomy. The remaining steps were as follows: A 0-Monocryl™ violet (poliglecaprone-25) or a 0-PDS-II (polydioxanone) suture with a 36-mm needle (Ethicon Inc., NJ, USA) was placed first on the right USL, proximal to the ischial spine and 1-3 cm away from its uterine insertion, then helically proceeded by 1 to 3 bite(s) (depending on the length of the ligament) for suspension/plication. The suture continued circumferentially in counter clockwise direction on the line between the cervicovaginal junction and the bladder in a full-thickness purse string fashion, at least 1 cm away to the bladder. This suture symmetrically ended in the left USL, with forming nearly an Ohm sign (Ω). Colpotomy was performed circumferentially using laparoscopic cold scissors and/or knife, maintaining a safe distance from the suture line. Following removal of the uterus, both ends of the prior suture line were knotted.
  Arms: Modified technique (MT)
Procedure: Standard technique (ST) — The conventional standard total laparoscopic hysterectomy technique was used in this control group.
  All operations were performed under general anaesthesia with nasogastric intubation and a bladder catheter in place. Cefazolin 2 g was administered to all patients for prophylaxis 30 min prior to surgery. Operations were performed with a 10-mm laparoscope (Karl Storz, Germany) through the trocar placed usually in the umbilicus. Two lateral 5-mm trocars and one midline 10-mm trocar were used. The placement of trocars varied according to the uterine size. Haemostasis was usually performed using bipolar forceps (Karl Storz Robi, Germany), whereas dissection was performed using the LigaSure™ (Covidien, Medtronic, USA). Maryland jaw laparoscopic sealer/divider, bipolar forceps and scissors. Colpotomy was performed with electrocautery devices and sutured intracorporeally.
  Arms: Standard technique (ST)

SUMMARY:
Modified Bakay technique offers a novel colpotomy and cuff closure technique for total laparoscopic hysterectomy (TLH), and consists of placing a single continuous running purse-string suture facilitating the cuff closure before colpotomy. The modified Bakay technique adds a standard apical compartment support and has the potential to facilitate the primary healing of the vaginal cuff. This study aimed to compare the surgical and clinical outcomes of the Modified Bakay technique to conventional standard technique in patients undergoing TLH.

DETAILED DESCRIPTION:
The basis for minimizing the rate of severe haemorrhage and ureteral injuries, the most serious events related to these steps, is meticulous dissection providing a clear operative field and the skill and experience of the surgeon. In total laparoscopic hysterectomy (TLH), the altered anatomy after the removal of the uterus may cause the retraction of vagina and shifting of neighbouring structures such as bladder and/or bowel to this pouch, thereby, leading to obstruction of the operative field for vaginal cuff closure.

Bakay published his novel colpotomy and cuff closure technique for TLH. It was the first to describe placing a single continuous running purse-string suture facilitating the cuff closure before colpotomy. The main advantage of the technique involved retrieving the safe suture margins required for vaginal cuff closure before the pelvic anatomy was altered by the removal of the uterus.

In addition to this advantage, we modified the technique to achieve a better cuff healing and standardized apical support and the modified Bakay technique (MT) proposes:

i) placing a single continuous running purse-string suture for vaginal cuff closure before the pelvic anatomy is altered by the colpotomy and removal of the uterus;

ii) suspension/plication of USLs (as a well-defined, efficient, concomitant apical support procedure to prevent future vaginal vault prolapse) routinely in each case before colpotomy while the margins of these ligaments and adjacent structures such as ureters are still prominent and pelvic anatomy is not altered; and

iii) using cold-knife colpotomy instead of electrosurgical colpotomy to support the primary healing of the vaginal cuff. In the present study, we aimed to compare the surgical and clinical outcomes of the MT to standard technique (ST) in patients undergoing TLH.

ELIGIBILITY:
Inclusion Criteria:

* Patients who needed laparoscopic hysterectomy

Exclusion Criteria:

* Patients with anaesthetic contraindications to laparoscopy
* premalignant or malignant genital disease
* prior pelvic and/or abdominal radiotherapy
* large adnexal masses; large fibroids obscuring the visualization of the cervicovaginal junction
* Suspicion of malignancy
* Pelvic organ prolapse Stage >2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Total operative time | Intraoperative, During the surgery
  Time interval between the placement and removal of primary trocar, as measured with minutes.
Surgical complications | During the surgery, at 7th, 30th and 90th day after the surgery.
  Intraoperative and postoperative complications related with the surgery. Any minor and major (e.g., bowel injury, bleeding>300cc, major vessel injury, bowel injury, haematoma, infection) complications will be classified according to the Clavien-Dindo classification system. This system allows to grade the adverse events between any deviation from the normal post-operative course not requiring surgical, endoscopic or radiological intervention (Grade 1), complications requiring drug treatments (Grade 2), Complications requiring surgical, endoscopic or radiological intervention (Grade 3), Life-threatening complications (Grade 4) and to the death of the patient (Grade 5).
Vaginal length | Postoperative, at 90th day after the surgery.
  The length of vagina from cervix to introitus, as measured with vaginal measuring ruler by cm.
Patient Satisfaction | Postoperative, at 90th day after the surgery.
  Patient satisfaction will be measured with Patient Global Impression of Improvement (PGI-I). It is scored as: Very much better (1), Much better (2), A little better (3), No change (4), A little worse (5), Much worse (6), Very much worse (7). Patient reported as Very much better or much better will be regarded as satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Kadir Bakay, Assoc Prof, Principal Investigator — Ondokuz Mayis Universitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Egemed Hospital, Aydin
  - Samsun Ondokuz Mayis University, Samsun

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon request from Uzeyir Kalkan (uzekal@hotmail.com).

REFERENCES:
- [Background] Bakay K. Introduction of a Novel Modification in Laparoscopic Hysterectomy: The Bakay Technique. J Minim Invasive Gynecol. 2018 Jul-Aug;25(5):916-919. doi: 10.1016/j.jmig.2018.03.013. Epub 2018 Mar 27. PMID 29602001
- [Derived] Kalkan U, Bakay K. A multimodal concept for vaginal cuff closure by modification of the Bakay technique in total laparoscopic hysterectomy: a randomized clinical study. BMC Womens Health. 2022 Jan 8;22(1):6. doi: 10.1186/s12905-021-01591-z. PMID 34996427